CLINICAL TRIAL: NCT04037007
Title: Efficacy and Safety of Precut Fistulotomy vs Conventional Cannulation Technique as a Primary Approach to Biliary Access According to the Endoscopist Experience Degree in ERCP
Brief Title: Efficacy of Fistulotomy for Biliary Cannulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2019-3601-147
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cholangiocarcinoma; Choledocholithiasis; Cholangitis; Pancreatic Cancer; Pancreatitis
Keywords: Precut sphincterotomy; Fistulotomy; Biliary cannulation; Efficacy
MeSH Terms: conditions — Cholangiocarcinoma; Choledocholithiasis; Cholangitis; Pancreatic Neoplasms; Pancreatitis | interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: We aim to perform a randomized clinical trial comparing fistulotomy (F) precut vs guidewire cannulation (CC), as a primary cannulation technique, and compare outcomes between high experienced endoscopists (> 200 ERCPs) and low experienced endoscopists (< 200 ERCPs).
Who Masked: Participant
Masking Description: The participant will be allocated to one group of the intervention conventional guidewire biliary cannulation or fistulotomy based on program software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fistulotomy - High experienced (Active Comparator): Fistulotomy precut with a needle knife, ERBE Endocut I, Effect 2; as the primary cannulation technique in high experienced endoscopists.
  Interventions: Procedure: Fistulotomy - High experienced.
- Fistulotomy - Low experienced (Active Comparator): Fistulotomy precut with a needle knife, ERBE Endocut I, Effect 2; as the primary cannulation technique in low experienced endoscopists.
  Interventions: Procedure: Fistulotomy - Low experienced.
- Conventional (guidewire) cannulation- High experience (Active Comparator): Conventional cannulation with an sphincterotome and 0.035 inch hydrophilic tip guidewire as the primary cannulation technique in high experienced endoscopists.
  Interventions: Procedure: Conventional (guidewire) cannulation- High experienced
- Conventional (guidewire) cannulation - Low experienced. (Active Comparator): Conventional cannulation with an sphincterotome and 0.035 inch hydrophilic tip guidewire as the primary cannulation technique in low experienced endoscopists.
  Interventions: Procedure: Conventional (guidewire) cannulation - Low experienced

INTERVENTIONS:
Procedure: Fistulotomy - High experienced. — We will perform a duodenoscopy, once located next to the papilla, we will perform precut fistulotomy on the papillary infundibulum with a needle knife with EBRE, EndoCut I, Effect 2, until biliary fluid exit is seen or the biliary duct is noted, then we will access to the biliary tree to complete de procedure.
  Arms: Fistulotomy - High experienced
Procedure: Fistulotomy - Low experienced. — We will perform a duodenoscopy, once located next to the papilla, we will perform precut fistulotomy on the papillary infundibulum with a needle knife with EBRE, EndoCut I, Effect 2, until biliary fluid exit is seen or the biliary duct is noted, then we will access to the biliary tree to complete de procedure.
  Arms: Fistulotomy - Low experienced
Procedure: Conventional (guidewire) cannulation- High experienced — We will perform a duodenoscopy, once located next to the papilla, we will perform cannulation with sphincterotome and hydrophilic tipped guidewire aided by fluoroscopy, once the guidewire reaches de common bile duct (seen on fluoroscopy) we will continue with the procedure according to the patient's indication.
  Arms: Conventional (guidewire) cannulation- High experience
Procedure: Conventional (guidewire) cannulation - Low experienced — We will perform a duodenoscopy, once located next to the papilla, we will perform cannulation with sphincterotome and hydrophilic tipped guidewire aided by fluoroscopy, once the guidewire reaches de common bile duct (seen on fluoroscopy) we will continue with the procedure according to the patient's indication.
  Arms: Conventional (guidewire) cannulation - Low experienced.

SUMMARY:
Access to the main bile duct is the first step in order to perform a therapeutic maneuver for biliary diseases. Early precut has been shown to ameliorate cannulation success rate, specially in difficult cannulation cases, when compared to guidewire cannulation (which is considered, for most, the standard technique). We aim to perform a randomized clinical trial comparing fistulotomy (F) precut vs guidewire cannulation (CC), as a primary cannulation technique, and compare outcomes between high experienced endoscopists (> 200 ERCPs[Endoscopic Retrograde cholangiopancreatography]) and low experienced endoscopists (< 200 ERCPs).

DETAILED DESCRIPTION:
Endoscopic Retrograde Pancreatography Cholangiography (ERCP) is the standard procedure for the treatment of pathologies that affect the bile duct. Approaching to the ampulla followed by deep selective biliary cannulation is the first step in order to apply any therapeutic method for bile duct pathologies. In patients with a normal anatomy it is estimated that about 11% of therapeutic ERCPs will be considered difficult biliary cannulation (duration of cannulation> 5 minutes, more than 5 attempts, > 1 cannulation of the main pancreatic duct). When early conventional precut has been compared to guidewire cannulation, cannulation success is in favor of precut with 86.7% compared to 66.7%; with a lower post-ERCP acute pancreatitis event rate: 6.1% vs 9.1%.

Objective: To determine the rate of biliary cannulation by comparing two techniques (fistulotomy versus standard biliary cannulation technique with guidewire) according to the endoscopist experience in ERCP.

Material and methods: A randomized prospective clinical trial will be conducted in the gastrointestinal endoscopy department of the CMN SXXI specialties hospital between the period of August 2019 and March 2020. 2 groups will be assigned as following: in group A the primary approach to access the bile duct will be conventional cannulation (CC) with guidewire, and group B for fistulotomy (F). On the other hand, there will be 2 groups of endoscopists (high experience> 200 ERCP) [HE] and low experience (<200 ERCP) [LE]. In total 4 groups: CCHE, CCLE, FHE, FLE. All patients undergoing ERCP with suspected or confirmed of choledocholithiasis, malignant and benign stenosis of the bile duct, men and women between 18 and 90 years will be included. Exclusion criteria: patients with previous ERCP, gastro-duodenal anatomy altered by previous surgery, suspicion or diagnosis of ampullary neoplasm, duodenal cancer, periampullar diverticula types 1 and 2, pregnant women, coagulopathy with INR greater than 1.5. Elimination criteria: patients with incomplete ERCP due to adverse anesthesia events. The reason and indication of the ERCP study will be determined, a data collection sheet will be used compiling: clinical data such as age, sex, concomitant diseases, symptoms, biochemical data, imaging studies (abdominal ultrasound, abdominal CT and MRCP), findings on ERCP (characteristics of the papilla, presence of periampullar diverticula); details of the cannulation technique such as the number of attempts, time to access the bile duct. A comparison will be made between both techniques and both groups HE and LE. The success rate of biliary cannulation and complication for both groups of doctors and maneuvers used will be documented.

Statistical analysis: Continuous variables will be described with mean, median or standard deviation according to their distribution; and categorical variables will be described as percentages. Categorical variables will be compared using Chi-square or Fisher's exact test, while quantitative variables will be compared using T-Student or Mann Whitney U test. A P less than 0.05 will be considered statistically significant (for T-Student and Mann-Whitney U will be 2-tailed). A sample size of 80 patients for each group was calculated.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing ERCP with suspected or confirmed of choledocholithiasis, malignant and benign biliary stenosis.

Exclusion Criteria:

* patients with previous ERCP, altered gastro-duodenal anatomy by previous surgery, suspicion or diagnosis of ampullary neoplasm, duodenal cancer, periampullary diverticula types 1 and 2, pregnant women, coagulopathy with INR greater than 1.5.

Elimination Criteria:

- Incomplete procedure due to anesthesia adverse events.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cannulation success rate within 5 minutes | 8 months
  Successful access to the main biliary duct and subsequently to the biliary tree

SECONDARY OUTCOMES:
Adverse event rate | 8 months
  Post-ERCP pancreatitis, perforation and bleeding rates
Technical success | 8 months
  Therapeutic success according to the patient indication

CONTACTS AND LOCATIONS:
Overall Officials: Oscar V Hernandez Mondragon, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Medico Nacional Siglo XXI Hospital de Especialidades, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopes L, Dinis-Ribeiro M, Rolanda C. Early precut fistulotomy for biliary access: time to change the paradigm of "the later, the better"? Gastrointest Endosc. 2014 Oct;80(4):634-641. doi: 10.1016/j.gie.2014.03.014. Epub 2014 May 6. PMID 24814775
- [Background] Jin YJ, Jeong S, Lee DH. Utility of needle-knife fistulotomy as an initial method of biliary cannulation to prevent post-ERCP pancreatitis in a highly selected at-risk group: a single-arm prospective feasibility study. Gastrointest Endosc. 2016 Nov;84(5):808-813. doi: 10.1016/j.gie.2016.04.011. Epub 2016 Apr 19. PMID 27102829
- [Background] Furuya CK, Sakai P, Marinho FRT, Otoch JP, Cheng S, Prudencio LL, de Moura EGH, Artifon ELA. Papillary fistulotomy vs conventional cannulation for endoscopic biliary access: A prospective randomized trial. World J Gastroenterol. 2018 Apr 28;24(16):1803-1811. doi: 10.3748/wjg.v24.i16.1803. PMID 29713133
- [Background] Abu-Hamda EM, Baron TH, Simmons DT, Petersen BT. A retrospective comparison of outcomes using three different precut needle knife techniques for biliary cannulation. J Clin Gastroenterol. 2005 Sep;39(8):717-21. doi: 10.1097/01.mcg.0000173928.82986.56. PMID 16082283
- [Background] Mavrogiannis C, Liatsos C, Romanos A, Petoumenos C, Nakos A, Karvountzis G. Needle-knife fistulotomy versus needle-knife precut papillotomy for the treatment of common bile duct stones. Gastrointest Endosc. 1999 Sep;50(3):334-9. doi: 10.1053/ge.1999.v50.98593. PMID 10462652